CLINICAL TRIAL: NCT04231994
Title: Prospective, Randomized, Single-center, Open-label, Parallel-group Trial Investigating the Efficacy of Therapeutic Plasma Exchange as an Adjunctive Strategy Against Early Septic Shock - Effect on Hemodynamics and Biochemical Markers
Brief Title: Therapeutic Plasmaexchange in Early Septic Shock
Acronym: EXCHANGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Stahl, Klaus Dr., Dr. Klaus Stahl, Fellow Gastroenterology and Critical Care Medicine, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXCHANGE 2786-2015
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Septic Shock
Keywords: Septic shock; Therapeutic plasma exchange; Sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPE (Experimental): additive singular therapeutic plasma Exchange (TPE) using fresh frozen Plasma (FFP) as replacement fluid
  Interventions: Device: TPE
- SMT (No Intervention): Standard medical Treatment (SMT) for septic shock following the present surviving sepsis guidelines

INTERVENTIONS:
Device: TPE — singular Therapeutic Plasma Exchange using fresh frozen Plasma as replacement fluid
  Arms: TPE

SUMMARY:
Sepsis is defined by the occurrence of critical organ dysfunction in the context of infection. Unfortunately, its incidence appears to be rising, and the mortality of septic shock remains extraordinary high (> 60%). Death in sepsis arises from shock and multi organ dysfunction that are - at least in part - triggered by an inadequate response of the host's immune system to the infection. Given the injurious role of 1) this overwhelming immune response and 2) the consumption of protective plasmatic factors (e.g. vWF cleaving proteases, hemostatic factors etc.) while the disease is progressing the investigators hypothesize that early therapeutic plasma exchange (TPE) in the most severely ill individuals might improve hemodynamics, oxygenation and ultimately survival. This therapeutic strategy combines 2 major aspects in 1 procedure: 1. removal of harmful circulating molecules and 2. replacement of protective plasma proteins. The investigators designed the EXCHANGE trial to analyze in a randomized fashion the benefit of TPE as an add-on treatment to state of the art standard sepsis care. Only patients with early septic shock (< 24 hrs) and high catecholamine doses (norepinephrine > 0.4 ug/kg body weight/min) will be included. Those in the treatment group will receive 1 TPE within 2 hours following randomization. The primary outcome is norepinephrine dose 6 hrs after randomization. The recruitment period is 2 years and will be performed at the Hannover medical School University hospital in Germany. Secondary endpoints (including organ dysfunction as well as biochemical markers of inflammation and coagulation) will be assessed on day 1-8 and day 28 after TPE.

The investigators hope to demonstrate a potential benefit of an additive treatment approach to improve the outcome of patients suffering from septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Onset of septic shock within less than 24 hrs
* Norepinephrine dose of ≥ 0.4 ug/kg/min bodyweight (target mean arterial pressure ≥ 65 mmHg) ≥ 30 min

Exclusion Criteria:

* Age<18 years and > 80 years
* Pregnancy
* Known history of transfusion reactions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Norepinephrine dose | 6 hours after randomization
  Vasopressor dose reduction as indicator of shock reversal

SECONDARY OUTCOMES:
Mean Sequential organ failure assessment (SOFA) score | day 1-8 following randomization
  SOFA score as indicator of organ dysfunction
percent change of ADAMTS-13 activity from baseline | 6 hours after randomization
  (will only be analyzed in the Hannover cohort)
percent change of activated Protein C activity from baseline | 6 hours after randomization
  (will only be analyzed in the Hannover cohort)
percent change of permeability factors angiopoietin-1, -2 and sTie-2 from baseline | 6 hours after randomization
  permeability and anti-permeability factors (will only be analyzed in the Hannover cohort)
28 day survival | after 28 days following randomization

CONTACTS AND LOCATIONS:
Overall Officials: Sascha David, MD, Principal Investigator — Clinic for nephrology; Klaus Stahl, MD, Principal Investigator — Clinic for gastroenterology and hepatology
Locations (2):
- Germany (2):
  - Hannover Medical School, Hanover, Lower Saxony
  - University Hospital Bonn, Bonn

IPD SHARING:
Plan to Share IPD: Yes
pre-defined substudies

REFERENCES:
- [Result] David S, Bode C, Putensen C, Welte T, Stahl K; EXCHANGE study group. Adjuvant therapeutic plasma exchange in septic shock. Intensive Care Med. 2021 Mar;47(3):352-354. doi: 10.1007/s00134-020-06339-1. Epub 2021 Jan 20. No abstract available. PMID 33471132
- [Derived] Stahl K, Wand P, Seeliger B, Wendel-Garcia PD, Schmidt JJ, Schmidt BMW, Sauer A, Lehmann F, Budde U, Busch M, Wiesner O, Welte T, Haller H, Wedemeyer H, Putensen C, Hoeper MM, Bode C, David S. Clinical and biochemical endpoints and predictors of response to plasma exchange in septic shock: results from a randomized controlled trial. Crit Care. 2022 May 12;26(1):134. doi: 10.1186/s13054-022-04003-2. PMID 35551628
- [Derived] Stahl K, Hillebrand UC, Kiyan Y, Seeliger B, Schmidt JJ, Schenk H, Pape T, Schmidt BMW, Welte T, Hoeper MM, Sauer A, Wygrecka M, Bode C, Wedemeyer H, Haller H, David S. Effects of therapeutic plasma exchange on the endothelial glycocalyx in septic shock. Intensive Care Med Exp. 2021 Nov 24;9(1):57. doi: 10.1186/s40635-021-00417-4. PMID 34817751
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33471132/